CLINICAL TRIAL: NCT03718689
Title: The Effect of Er:YAG Laser on Clinical Success of a Hydrophilic Fissure Sealant
Brief Title: Effect of Er:YAG Laser on Hydrophilic Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-048
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Fissure Sealant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group L (Experimental): The second group of teeth (Group L) were etched with Er:YAG laser.
  Interventions: Device: Laser etching
- Group A+L (Experimental): The third group of teeth (Group A+L) were etched with both Er:YAG laser and phosphoric acid.
  Interventions: Device: Laser etching
- Group A (No Intervention): The first group of teeth (Group A) were not etched with Er:YAG laser.

INTERVENTIONS:
Device: Laser etching — Acid etching
  Other Names: Acid
  Arms: Group A+L; Group L

SUMMARY:
This study was conducted on 44 (19 girls and 25 boys) patients presenting 132 permanent first molars, who applied for oral examination to Adnan Menderes University Faculty of Dentistry Department of Pediatric Dentistry. The patients involved in the study were aged between 7-11 years who had fully erupted permanent first molars, which were suitable for non-invasive fissure sealant application (narrow, deep fissures).

DETAILED DESCRIPTION:
The permanent first molar teeth were cleaned using a polishing brush and pumice and isolated with cotton rolls. Caries status was assessed using DIAGNOdent pen (DIAGNOdent pen 2190, KaVo, Biberach, Germany) at the occlusal and proximal sites. Teeth having DIAGNOdent readings of 12 or less at the occlusal site and 7 or less at the proximal site were included in the study. Then, the teeth were divided into three groups. The first group (Grup A) of teeth were etched with phosphoric acid, the second group of teeth (Group L) were etched with Er:YAG laser and the third group of teeth (Group A+L) were etched with both Er:YAG laser and phosphoric acid. The patients were recalled for follow up examination at the 3rd, 6th and 9th months. The teeth were assessed using mouth mirror and explorer regarding new caries formation and retention of the fissure sealants. The obtained data were analyzed using SPSS 24.0 (SPSS 24.0 for Windows, SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in this study had good general health and oral hygiene.
* Fully erupted permanent first molar teeth with deep, narrow fissures
* Teeth with no detectable occlusal and proximal caries

Exclusion Criteria:

* Hypomineralized areas such as fluorosis, molar incisor hypomineralization
* Allergy to resins, who were not willing to participate in the study.
* Teeth with hypomineralized areas such as fluorosis,
* Teeth with molar incisor hypomineralization

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Retention rate | Change from Baseline retention rate at 12 months
  Clinical success

CONTACTS AND LOCATIONS:
Locations (1):
- Hülya Yılmaz, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The results will be shared with other researchers.

REFERENCES:
- [Result] Guclu ZA, Hurt AP, Donmez N, Coleman NJ. Effect of Er:YAG laser enamel conditioning and moisture on the microleakage of a hydrophilic sealant. Odontology. 2018 Jul;106(3):225-231. doi: 10.1007/s10266-017-0323-4. Epub 2017 Dec 13. PMID 29236177